### UNIVERSITY OF SOUTH CAROLINA CONSENT TO PARTICIPATE IN A RESEARCH STUDY

## Importance of Summer Day Camps on Child Health

Dear Parent or Guardian,

Your child is invited to participate in a study being conducted by Glenn Weaver. I am a Professor in the Arnold School of Public Health, at the University of South Carolina. The study also involves obtaining information from you about your child and yourself.

The University of South Carolina, Department of Exercise Science and the National Institutes of Health are sponsoring this research study.

This form explains what is involved. We would like you to read it closely and ask any questions that you have before you decide to let your child participate.

Your child is invited to participate because he/she will be in kindergarten-4<sup>th</sup> grade and the Boys & Girls Club of the Upstate offers a summer camp at his/her school

The following is a short summary of this study to help you decide whether to be a part of this study. More detailed information is listed later in this form.

Please keep this letter for your records and in case you have future questions.

#### **KEY INFORMATION ABOUT THIS STUDY**

#### WHAT IS THE PURPOSE OF THIS STUDY?

Attending a summer camp has the potential to impact children's health behaviors like physical activity, diet, sleep, and screen time in a positive way. In turn attendance could stop children from gaining unhealthy weight during the summer. However, many families do not have the resources to send their children to summer camps. The purpose of this project is to understand if providing a voucher to attend 8 weeks of a summer day camp will increase children's attendance at a summer day camp in comparison to children who do not receive a voucher to attend a summer camp. We will also examine the health benefits children receive from attending a summer day camp in comparison to children that do not attend a summer camp. This information is important to help develop community-based programs for children outside of school.

| 1 year – end of school year (spring—2 weeks), summer, and start of school year (fall), spring |
|---|
| ur school, parents, and children to do? |
| Students wear physical activity FitBit-like device for 2 weeks during school and again during summer |
| Measure height and weight at the end and beginning of the school year |
| Parents complete <b>brief survey</b> about your child, their physical activity, screen-time, sleep, dietary behaviors, and other related behaviors (<30min) – survey is sent via text to parent's smartphones (school and summer) |
| Parents complete <b>10 daily diaries</b> (<5min each) in the evenings during the 2-weeks. Diaries ask about what the child did that day - survey is sent via text to parent's smartphones (school and summer) |
| There are no foreseeable risks involved for parents of children for participating in this study. All information will remain confidential. |
| We will use this information to work with schools and other community partners in designing programs that help children lead healthy lives when they are away from school |

#### WHAT WILL HAPPEN DURING THIS STUDY?

If you agree your child will be **randomly assigned** to one of four groups.

You do not have a choice about which group your child joins.

- 1. <u>Group 1</u> children in this group receive a voucher to cover the cost of attending a summer day camp for 8 weeks FREE of charge. Additionally, these children will wear a Fitbit device during the summer and parents will receive weekly updates about their child's sleep and physical activity. Finally, children will meet with the research staff on several occasions during the year to be weighed, measured and complete other evaluations
- 2. **Group 2** children in this group receive a voucher to cover the cost of attending a summer day camp for 8 weeks FREE of charge as well as meeting with the research staff on several occasions during the year to be weighed, measured and complete other evaluations.
- 3. **Group 3** children will wear a Fitbit device during the summer and parents will receive weekly updates about their child's sleep and physical activity as well as meeting with the research staff on several occasions during the year to be weighed, measured and complete other evaluations.
- 4. **Group 4** children in this group will meet with the research staff the same as those in Group 1. Instead of a voucher, children in the group are eligible to receive gift cards up to \$100 worth for each visit they complete.

If more families agree to participate than we can accommodate we will randomly select families to participate in the study.

Twice during the year (spring semester and summer vacation) your child will wear a wristwatch activity monitor, like a FitBit, for 14 days. After completing the 14 days, the monitor will be returned to the research team.

During your child's PE class at the beginning and end of the school year as well as the beginning of the next school year, your child's height and weight will measured.

At each school and summer visit, we will ask that you, the parent/guardian of the child, complete a series of questions related to:

- Your child's dietary intake and physical activity
- Any rules you have regarding your child's food and activity
- How much screen time, such as TV, video games, and computer, your child uses
- Complete 14 daily diaries of your child's bed time and when they wake up

For the summer measurements, we will hold multiple day-long events on the weekends at your child's school. We will notify you by TEXT of the dates and provide free food and drinks to everyone that arrives to pick up their wrist-watch and complete the questionnaires.

#### **HOW LONG WILL IT TAKE?**

Each parent/child will participate for one year.

| Fall School<br>(August/Sept) | Spring School<br>(April/May) | Summer<br>(June/July) | Fall School<br>(August/Sept) |
|---|---|---|---|
| Height and Weight<br>Measured during PE | Height and Weight Measured during PE | Summer Day Camp<br>OR | Height and Weight<br>Measured during PE |
| Amount of time: ~2 minutes | Amount of time: ~2 minutes | Comparison group | Amount of time: ~2 minutes |
| | 2 Weeks - Child wears Fitbit-<br>like device and Parent<br>completes short surveys on<br>smartphone | 2 Weeks - Child wears Fitbit-like device and Parent completes short surveys on smartphone | |
| | Amount of time: Device placement <2 minutes, Parent surveys 30-45 minutes | Amount of time: Device placement <2 minutes, Parent surveys 30- 45 minutes | |

Completing all survey questions will take 30 to 45 minutes during school and again during summer.

#### WILL I BE PAID FOR PARTICIPATING?

If your child is assigned to Group 3 or 4, you will receive up to \$100 for attending visits, completing questionnaires, diaries and interviews. Payments will be distributed as \$25 for completing school year measures and \$75 for completing summer measures. Payment will be in the form of an electronic Amazon gift card sent via TEXT.

If your child is assigned to Group 1 or 2, you will receive a voucher to cover the cost of eight weeks of summer camp for your child.

#### WHAT ARE THE RISKS OF THIS STUDY?

There are no foreseeable risks associated with participating in this study.

There are no additional risks in attending the summer day camp. For children, the risk to wearing the wrist-placed activity monitor is minimal. The monitor is easily placed on the wrist and worn much like a wristwatch. The monitor is water proof and can be worn during showering but should be removed during baths and swimming.

The surveys focus exclusively on your role in terms of your child's eating and physical activity. You may leave blank any sections of the questionnaire that you do not wish to complete. While all precautions will be taken to ensure your privacy, there is a chance that your privacy/confidentiality may be breached. If this occurs, we will notify you of the breach and take any necessary steps to remedy the situation.

#### WHAT ARE THE BENEFITS OF THIS STUDY?

We believe the potential benefits will be a greater understanding of the influence of summer programming on the health outcomes of children and what occurs during the summer and how this leads to accelerated weight gain. From this information, we will work with the schools and other community entities serving children outside the regular school day to develop opportunities that help children maintain a healthy weight over summer vacation.

#### WILL IT COST ANYTHING TO PARTICIPATE?

There will be no costs to you for participating in this study other than possible costs related to transportation to and from the school sites in the summer to pick-up/drop-off data collection materials.

#### DO I HAVE A CHOICE TO BE IN THE STUDY?

Children and parents/guardians are free to withdraw consent and discontinue participation in the study at any time without penalty or loss of benefits. Your decision of whether to let your child participate is not connected with his/her school work and not participating will not impact his/her standing with the school.

There is no penalty for not participating.

Participants may withdraw from the study at any time without penalty.

The school district is neither sponsoring nor conducting this research.

#### WHO WILL SEE THE INFORMATION I GIVE?

All data collected during this study is strictly confidential. No data will be looked at by anyone other than the university research staff. Parents and/or guardians will not be informed of their child's responses to any of the survey answers, nor will children be informed of their parent/guardian's responses. Data will be stored in locked filing cabinets and protected computer files at the University of South Carolina. Participants will never be identified in any reports, papers, or publications coming from this study. A participant ID number will be assigned to each child and family at the beginning of the study and this number will be used for record keeping and data analysis. Your/your child's information collected as part of the research study will not be used or distributed for future research studies.

#### **VOLUNTARY PARTICIPATION**

Participation in this research study is voluntary. You are free not to participate, or to stop participating at any time, for any reason without negative consequences. If you do withdraw from this study, the information you have already provided will be kept in a confidential manner. If you wish to withdraw from the study, please call or email the principal investigator listed on this form.

#### **CLINICAL TRIAL REGISTRY DATABANK**

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

#### NOTIFICATION OF PARTICIPATION

We will notify parents/children via TEXT of their participation in the study within one month of receiving the signed form at the end of this document.

In the event more parents/children want to participate than the project can accommodate, we will randomly select parents/children to take part in the study.

#### WHAT IF I HAVE QUESTIONS ABOUT THIS STUDY?

If you have any questions, please call:

Name: Emily Tyler, Project Coordinator

Phone/TEXT: 803-429-0320

Email: **HealthySummerStudy@gmail.com** 

Questions about your rights as a research subject are to be directed to:

Lisa Johnson, Assistant Director
Office of Research Compliance, University of South Carolina
1600 Hampton Street, Suite 414D
Columbia, SC 29208
Phone: (803) 777-7095 or email: LisaJ@mailbox.sc.edu

Please keep this letter for your records and in case you have future questions.

If you wish to participate, please sign and complete the form below

# Importance of Summer Day Camps PLEASE RETURN THIS SHEET TO YOUR CHILD'S PE CLASS

I have read and understand the description of this study and what will happen during. I have been given opportunity to ask questions about participation in this study and I have received a copy of this informed consent form to keep.

#### Please check one of the following:

| YES I agree to my child's and n | I agree to my child's and my participation in the study |
|---|---|
| NO I do not agree to my child's and my participation in the study | |
| Parent/Guardian's Signature | Date |
| Parents/Guardian's PRINTED First and Last NAME | Your Relationship to the Child (Mother, Father, Grandma, etc) |
| Child's PRINTED First and Last Name | Child's Date of Birth<br>(mm/dd/yyyy) |
| If "YES", please include your <u>contact information</u> and complete questions on the next page | |
| Your Street Address City, Zip | |
| ( ) | ( ) |
| Your Primary Cell Phone Number (555)555-5555 | Alternate Cell Phone Number (555)555-5555 |
| Your Email Address | Alternate Email Address |

### IF "YES", PLEASE COMPLETE THE FOLLOWING INFORMATION

| WHAT IS THE HIGHEST LEVEL OF EDUCATION YOU HAVE COMPLETED? | |
|---|---|
| Less than High School | High School |
| Some College or Vocational Training | Completed College or University |
| Completed Graduate or Professional Degree | |
| WHAT IS <u>YOUR CHILD'S</u> GRADE? | |
| Kindergarten 1 <sup>st</sup> Grade | 2 <sup>nd</sup> Grade |
| 3 <sup>rd</sup> Grade 4 <sup>th</sup> Grade | 5 <sup>th</sup> Grade |
| WHAT IS YOUR CHILD'S <u>GENDER</u> ? (circle one) | Boy Girl |
| PLEASE INDICATE IF <u>YOU USE</u> ANY OF THE FOLLOWI | NG: Yes, No, I do not use. |
| WIC (Women, Infants, and Children) | |
| SNAP (Supplemental Nutrition Assistance Program) | |
| Covered by <b>Medicaid</b> Insurance | |

**Luther Vaughan**